CLINICAL TRIAL: NCT02179879
Title: Protocol for Development and Validation of Metrics for Conventional Lumbar Epidural Catheter Placement for Labor Analgesia in Obstetric Patients
Brief Title: Development and Validation of Metrics Lumbar Labor Epidural Catheter Placement
Status: Completed | Type: Observational
Sponsor: Cork University Hospital (Other)
Responsible Party: Principal Investigator, Karthikeyan Kallidaikurichi Srinivasan, Specialist Registrar,Anaesthetics,Cork University Hospital, Cork University Hospital
Other Study IDs: ECM4(U)01/10/13
Record Dates: First submitted 2014-06-30; First posted 2014-07-02 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Labor Pain
Keywords: labor,epidural,analgesia
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Video validation group: This will include video taping of experts (defined as one who has performed more than 500 labor epidurals in preceding 5 year period) and novices (defined as one who has done less than 50 epidurals in preceeding 2 years) perfoming labor epidural
  Interventions: Other: Video validation

INTERVENTIONS:
Other: Video validation — Video taping of anaesthetist (experts and novices) perfoming labor epidural.

SUMMARY:
Procedural skills play an important role in anaesthetic expertise. More focused training and assessment of procedural skills will be needed in the future as training moves from an apprenticeship based training system to competency based assessment.

Currently various techniques exists to assess procedural skills of anaesthetist. For epidural catheter placement, task specific check list, global rating scales and cumulative sum techniques have been developed and validated. These techniques aim either for better qualitative outcome sacrificing objectivity or rely on self-reporting. A decrease in objectivity in turn hampers inter-rater reliability which is an essential component of a valid assessment model. Checklists type assessments force the developer to comprehensively characterize the procedure of interest and then validate the completed procedure characterization. This approach has been quantitatively shown to have higher assessment reliability levels compared to Likert-scale assessment.

The objective of the project is to develop and validate a comprehensive procedure characterization for labor epidural catheter placement. Another objective is to compare this new assessment tool with existing checklist and global rating scale for labor epidural to establish concurrent validity.5 A well-developed objective, validated procedure characterization serves as a master tool which has multiple applications. It helps to build a training programme for the procedure, allows providing metrics based feedback to trainees using simulator, helps to assess the performance of trainees and in future might be used as benchmark to allow competency based progression in the training.

DETAILED DESCRIPTION:
Study part 1 After ethics committee approval a group of experts (n = 3 ) in conventional lumbar epidural catheter placement will be selected (an expert is defined as one who has performed more than 500 labor epidurals in preceding 5 year period). During a number of face-to-face meetings experts will identify, characterize and define the procedure. They will analyze task and identify units of behavior to be measured which constitute in a step-wise fashion how the procedure is optimally performed and deviations from optimal procedure performance as described previously. After informed consent from the patient and the anaesthetist performing the procedure, 2 video recordings of experts performing epidural and 2 video recordings of novices (defined as one who has done less than 50 epidurals) performing epidural will be recorded for detailed review during metric development meetings.

Study part 2 The developed metrics will be subjected to assessments of construct validity (a set of procedures for evaluating a testing instrument based on a degree to which the test terms identify the quality, ability or trait it was designed to measure) and concurrent validity (the evaluation in which the relationship between the test scores and the scores on the another instrument purporting to measure the same construct are related). We will also evaluated the inter-rater reliability of the metrics using i) proportion of agreement between raters, ii) correlation strength (using Pearson's Correlation Coefficient) and iii) Coefficient Alpha. After informed consent,10 experts (who are not a part of committee developing the metrics) each performing one or more lumbar epidural catheter placements for labor and 10 novices each performing one or more lumbar epidural catheter placements for labor will be video recorded. Two experts will review the video recording and score the performance based on checklist based system developed and compare with likert-scale checklists/global rating scale system.

ELIGIBILITY:
Inclusion Criteria:

* an expert is defined as one who has performed more than 500 labor epidurals in preceding 5 year period
* novice (defined as one who has done less than 50 epidurals in previous 2 years)

Exclusion Criteria:

* Non consenting anaesthetist
* Patients not consenting for video recording

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Expertes and novice anaesthetist perfoming labor epidural analgesia
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Construct validitiy | WIthin 12 months post recording epidural procedure video
  a set of procedures for evaluating a testing instrument based on a degree to which the test terms identify the quality, ability or trait it was designed to measure.In our study we aim to see if the metrics developed will be able to differentiate between experts and novices in performing the porcedure

SECONDARY OUTCOMES:
Concurrrent validity | within 12 months following completion of epidural video recording
  Concurrent validity is defined as a set of procedures for evaluating a testing instrument based on a degree to which the test terms identify the quality, ability or trait it was designed to measure.We aim to compare the interrater reliability of the metrics with compare with likert-scale checklists/global rating scale system developed already for the procedure.
Interrater reliability | 12 months from time of aquiring the epidural video
  We will evaluate the inter-rater reliability of the metrics using i) proportion of agreement between raters, ii) correlation strength (using Pearson's Correlation Coefficient) and iii) Coefficient Alpha

CONTACTS AND LOCATIONS:
Overall Officials: Karthikeyan Kallidaikurichi Srinivasan, FCARCSI,MD, Principal Investigator — Cork University Hospital
Locations (1):
- Cork University Hospital, Cork,Ireland, Ireland

REFERENCES:
- [Derived] Kallidaikurichi Srinivasan K, Gallagher A, O'Brien N, Sudir V, Barrett N, O'Connor R, Holt F, Lee P, O'Donnell B, Shorten G. Proficiency-based progression training: an 'end to end' model for decreasing error applied to achievement of effective epidural analgesia during labour: a randomised control study. BMJ Open. 2018 Oct 15;8(10):e020099. doi: 10.1136/bmjopen-2017-020099. PMID 30327396